CLINICAL TRIAL: NCT01165840
Title: Population Pharmacokinetic Analysis of Dapsone in Normal, Overweight and Obese Volunteers
Brief Title: Effect of Weight and/or Obesity on Dapsone Drug Concentrations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Ron Hall, Associate Professor, Texas Tech University Health Sciences Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMAIRB97; 5UL1RR024982-02 (NIH)
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Obesity; Leprosy; Tuberculosis
Keywords: Obesity; Pharmacokinetics; Dapsone; Leprosy; Tuberculosis
MeSH Terms: conditions — Obesity; Leprosy; Tuberculosis | interventions — Dapsone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dapsone (Experimental): Dapsone 100 mg PO x 1 dose
  Interventions: Drug: Dapsone

INTERVENTIONS:
Drug: Dapsone — 100 mg PO x 1 dose

SUMMARY:
This study will find how weight affects the dosing of a drug called dapsone. Currently, the amount of dapsone a patient receives is the same regardless of the patient's weight.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age >18 years, of all racial and ethnic origins.
* Non-English speaking Spanish speakers will be included in the study.
* We are recruiting 12 normal or underweight (BMI <25 kg/m2), 12 overweight or obese (BMI 25-40 kg/m2), and 12 extremely obese (BMI > 40 kg/m2) for this study. This index is calculated using the volunteer's height and weight (Formula: weight (lb) / [height (in)]2 x 703). Half of each group will be male; the other half will be female.

Exclusion Criteria:

* Pregnant or nursing or unwilling to use a reliable contraception method during the study. The effects of dapsone on pregnancy are unknown. In addition, the metabolic changes that accompany pregnancy may alter the concentration-time profile of dapsone, so that the pregnancy and post-partum state would be a confounding variable.
* Abnormal liver function tests: transaminases>10 times upper limit of normal, Alkaline phosphatase>5 times upper limit of normal, total bilirubin>5 times upper limit of normal.
* History of allergies to dapsone, sulfones, or sulfonamides.
* Dapsone, sulfones, or sulfonamides are contraindicated for any reason.
* Volunteers unwilling to comply with study procedures.
* Current suspected or documented infection of any kind.
* Volunteers with colon resection, gastric bypass, lap band, or any other conditions inhibiting gastric absorption of drug.
* Current or previous participation within 28 days of enrollment in another research study that involves the use of medication, contrast, or any other compound that may alter blood count and/or blood chemistry (liver function, kidney function or electrolyte balance), unless waved by PI.
* Donation of 450 milliliters (ml) (one unit) of blood or more within 8 weeks (56 days) prior to study enrollment, unless waved by PI.
* Current use of zidovudine, amprenavir, rifabutin, rifapentine, or saquinavir.
* Creatinine clearance < 70 ml/minute (min) as estimated by the Cockcroft-gault equation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hall, PharmD, MSCS, Principal Investigator — Texas Tech UHSC
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited into three BMI groups to ensure a wide total body weight distribution, but only one pharmacokinetic model was analyzed with total body weight being one of the potential covariates that was assessed.
Pre-assignment Details: Thirty-seven patient provided consent, but only 36 started the study. One patient provided informed consent but was found to have G6PD and was not allowed to continue.
Period: Overall Study
Arm/Group | Dapsone
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dapsone
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 34
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Serum Clearance
Description: Serum clearance of dapsone
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Dapsone
Number analyzed (Participants) | 36
L/h | 2.55 (1.24)

ADVERSE EVENTS:
Time Frame: 72 hours
Description: Participants were in the Clinical Research Unit under nursing supervision 0-24 hours after the dapsone dose. Research clinic visits occured at 48 and 72 hours after the dapsone dose under supervision of a research coordinator.
Arm/Group | Dapsone
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No